CLINICAL TRIAL: NCT06459011
Title: TAKINGCARE - TAcKlING the Needs of Carers of People With Chronic respirAtoRy disEases
Status: Recruiting | Type: Observational
Sponsor: Aveiro University (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Alda Sofia Pires de Dias Marques, Senior Lecturer, Aveiro University
Other Study IDs: PRT/BD/154726/2023
Record Dates: First submitted 2024-06-09; First posted 2024-06-14 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Chronic Respiratory Disease
Keywords: chronic respiratory disease; needs; informal care; loved ones; health literacy; measurement properties; preparedness for caregiving

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to: i) develop an instrument that assesses the needs of informal carers of people with chronic respiratory diseases (CRD), along diseases' trajectory, and evaluate its measurement properties; ii) identify existing instruments that assess the needs of informal/family carers and their measurement properties, iii) characterize the needs of informal carers of people with CRD and iv) characterize the health literacy of informal carers of people with CRD.

The first task will be a systematic review. For the second and third tasks, people with CRD, their informal carers and health professionals will be recruited via the pulmonology services from the hospitals:Unidade Local de Saúde de Gaia/Espinho, Unidade Local de Saúde da Região de Aveiro, and Unidade Local de Saúde de Entre o Douro e Vouga. On task 2, a mixed-methods study will be conducted to characterize the needs of informal carers of people with CRD, as well as their health literacy. On task 3, an instrument that assesses the needs of informal carers of people with CRD will be developed and its measurement properties will be studied.

This study is urgently needed to provide meaningful support to this hidden workforce who provides most of the care to people with DRC contributing to guide meaningful supportive care to this population and their loved ones.

DETAILED DESCRIPTION:
Chronic respiratory diseases (CRD) are the 3rd leading cause of death and disability worldwide, with high burden for individuals, but also for their families and society, including health services. They are systemic, with pulmonary and extrapulmonary manisfestations, and are characterized by a progressive decline on multiple activities of daily living making this people depend on others along diseases' trajectory.

Daily, informal/family carers, who may be relatives, partners, friends or neighbours, with a significant personal relationship with an elderly person or an adult with a disabling chronic disease, are the main source of support of people with CRD. They have a multiplicity of roles in providing physical, financial, psychological/emotional, social, and spiritual support. It is assumed that informal/family carers have the appropriate level of health literacy, disease knowledge, financial security, household conditions, psychological readiness, and medical care abilities to support the person with CRD.

Although they report positive experiences (e.g., personal growth, satisfaction), there has been an acknowledgement of negative impacts (e.g., burden, difficulty in realizing personal interests/projects) and specific needs related to their roles. Nevertheless, their needs are usually unmet and rarely assessed, and they are highly neglected by the social/health system, as well as in research. Assessment of this needs is the first step to provide meaningful support to this hidden workforce who provides most of the care to people with CRD and it has been emphasised by the European Union's recommendations to support and empower informal carers. However, only two instruments have been explicitly designed to assess their needs: the Carers' Alert Thermometer and the Carer Support Needs Assessment Tool (CSNAT), but their routine use is limited, their measurement properties have been scarcely explored and only for COPD, and studies have focused on end-of-life situations.

Therefore, the primary aim of this study is to develop a new instrument to assess the needs of loved ones across CRD' trajectory. Secondary aims are to map available instruments that assess the needs of informal/family carers and their measurement properties, and characterize the needs of informal carers of people with CRD and their health literacy.

This study will be carried out at the University of Aveiro, at the Laboratory of Research and Respiratory Rehabilitation of the School of Health Sciences of the University of Aveiro, at Unidade Local de Saúde de Gaia/Espinho, at Unidade Local de Saúde da Região de Aveiro, and at Unidade Local de Saúde de Entre o Douro e Vouga, in Portugal.

It comprises three tasks: task 1 will consist of a systematic review, in which the instruments that assess the needs of informal/family carers and their measurement properties will be identified; task 2 will be a cross-sectional study where the needs of informal carers of people with CRD and their health literacy will be characterized, through a mixed-methods study, integrating people with CRD, their informal carers, and health professionals; task 3 will be the development of an instrument that assesses the needs of informal carers of people with CRD. The items will be generated based on tasks 1 and 2 and following existing guidelines. The instrument will be pilot-tested, and the measurement properties of the instrument will then be tested in a cross-sectional observational study. On task 2, the Carer Support Needs Assessment Tool v3.0 and the Preparedness for Caregiving Scale will also be translated to European Portuguese.

Adults who are diagnosed with CRD, who are fluent in Portuguese and identify an informal/family carer will be included. If they show signs of cognitive impairment, they will not be eligible for the interviews. Informal carers will be included in the study if they are ≥18 years old and are fluent in Portuguese. They will be excluded if they show signs of cognitive impairment. Health professionals will be included if they contact with people with CRD in their clinical practice.

Sociodemographic and general clinical data will be collected. Instruments assessing cognitive impairment, functional capacity, disease's impact, health related quality of life, health status, level of anxiety and depression, satisfaction with life, social network, functionality, burden, positive aspects of caregiving, preparedness for caregiving, health literacy and informal carers' needs, as well as questions regarding care, will be applied. Interviews will be conducted.

Sample size will be determined by the saturation of qualitative data in task 2. For the assessment of health literacy of informal carers of people with CRD, it is not possible to determine the sample number. The maximum number of informal carers will be recruited and estimates a posteriori will be made. For task 3, following the Consensus-based Standards guidelines for the Selection of health status Measurement Instruments (COSMIN), a minimum of 100 participants will be required.

Data analysis will be conducted using the Statistical Package for the Social Sciences (SPSS) software. For the organization and visualization/analysis of qualitative data, the NVivo program will be used. Descriptive statistics, comparison of distributions, and associations. Validity and reliability will be assessed. The analysis of qualitative data will be divided into content analysis and thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* People with chronic respiratory diseases (CRD):

  * 18 years of age or older;
  * Diagnosed with ILD, COPD, lung cancer, severe asthma or bronchiectasis;
  * Fluent in Portuguese;
  * Identify an informal/family carer;
* Informal carers of people with CRD:

  * 18 years of age or older;
  * Fluent in Portuguese.
* Health Professionals:

  * Fluent in Portuguese;
  * Contact with people with CRD in their clinical practice.

Exclusion Criteria:

* People with CRD:

  * Signs of cognitive impairment in the Six-item Cognitive Impairment Test (6CIT) for the interviews.
* Informal carers of people with CRD:

  * Signs of cognitive impairment in the 6CIT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with chronic respiratory diseases, informal carers of people with chronic respiratory diseases, and health professionals
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Preparedness for Caregiving Scale (PCS) | Task 2 and 3 (baseline)
  The PCS was developed to assess the competence/level of preparation of informal/family carers (family member or friend) of elderly people with moderate to severe cognitive or physical decline at home.The scale has 8 items, scored on a 5-point scale (from 0 - "not at all prepared" to 4 - "very well prepared"). The total score varies from 0 to 32, with a higher score corresponding to a better perception of level of preparation It has shown good measurement properties. It will be translated and culturally adapted and applied to informal carers of people with CRD.

SECONDARY OUTCOMES:
Six Minute Walk Test (6MWT) | Task 2 and 3 (baseline)
  The 6MWT is the gold standard exercise test and is commonly used to assess functional status.It is a valid and reliable measure in CRD. It will be used to characterize participants with CRD.
: Chronic Airways Assessment Test (CAAT) | Task 2 and 3 (baseline)
  CAAT is a change to the COPD Assessment Test (CAT) so that it can be applied to people with COPD and/or asthma.It assesses diseases' impact, presenting 8 items related to respiratory symptoms (cough, chest symptoms and impacts on well-being and day-to-day, related to dyspnea, activity limitation, confidence to leave home, sleep and energy level), classified from 0 to 5. The total score is calculated by adding the score of the 8 items, ranging from 0 to 40 points, with a higher score corresponding to a greater impact of the disease. The total score can be divided into 4 levels: 1) low, 2) moderate, 3) high and 4) very high impact. The CAAT proved to be valid and reliable for people with COPD and/or asthma. Similarly, the CAT is a valid and reliable instrument, capable of discriminating people with different degrees of severity of COPD and has been used in different CRD. It will be used to characterize participants with CRD.
King's Brief Interstitial Lung Disease (KBILD) | Task 2 and 3 (baseline)
  The KBILD was the first questionnaire developed to evaluate health related quality of life (HRQoL) in adults with insterstitial lung disease (ILD). It is easy to administer/ (5 to 7 minutes), economic and with excellent measurement properties. It consists of 15 items with a Likert scale of 7 points [1 - always 7 - never (items 1, 2, 3, 4, 6, 14); 1 - never 7 - always (item 5); 1 - significantly 7 - not at all (item 15)]. The total score and/or the score by domain (psychological, dyspnoea and activities, and chest symtpoms) can be calculated. The scores are transformed logarithmically, ranging from 0 to 100, and a higher score corresponds to a better perception of HRQoL. It will be used to characterize participants with ILD.
5-level EuroQoL-5D (EQ-5D-5L) | Task 2 and 3 (baseline)
  The EQ-5D-5L was developed by the EuroQol group to assess the perception of a person's current health status. It includes 5 dimensions (mobility, personal care, usual activities, pain, anxiety/depression) with 5 response levels (no problems, mild, moderate, severe or extreme problems). It also includes a vertical visual analogue scale (EQ VAS), which quantifies the perception of health status, ranging from 0 ("the worst health you can imagine") to 100 ("the best health you can imagine"). Its score can be transformed into Quality Adjusted Life Years and used for cost-utility analyses. The EQ-5D-5L is a simple to use, valid, reliable and responsive measure. It will be applied to people with CRD and their informal carers.
Hospital Anxiety and Depression Scale (HADS) | Task 2 and 3 (baseline)
  The HADS was developed with the aim of providing health professionals with a reliable, valid and easy-to-use measure to identify and quantify the level of depression and anxiety.It consists of two subscales, which are scored separately: one for anxiety (seven items) and one for depression (seven items). Each item is scored from 0 to 3 points, so each subscale varies between 0 and 21 points. A score between 0 and 7 is 'normal', between 8 and 10 shows "light" level, between 11 and 14 "moderate" level, and between 15 and 21 "severe" level of anxiety/depression. It will be applied to people with CRD and their informal carers.
Satisfaction with life scale (SWLS) | Task 2 and 3 (baseline)
  The SWLS was developed to measure overall satisfaction with life as a cognitive component of well-being. The scale presents 5 items, scored from 1 (totally disagrees) to 7 (totally agrees), and the score varies from 5 to 35, with a higher score corresponding to a greater satisfaction with life. It is a widely used instrument and is valid, reliable and can be used in different age groups. It will be applied to people with CRD and their informal carers.
Lubben Social Network Scale - 6 items (LSNS-6) | Task 2 and 3 (baseline)
  The LSNS-6 is a reduced version of the Lubben Scale of Social Networks, which was developed for the assessment of social networks in the elderly population. The score varies from 0 to 30, and a higher score corresponds to a greater social network. A score of less than 12 corresponds to social isolation. It is used internationally and is valid and reliable. It will be applied to people with CRD and their informal carers.
World Health Organization Disability Assessment Schedule (WHODAS 2.0) | Task 2 and 3 (baseline)
  The WHODAS 2.0 was developed by the World Health Organization as a general measure of functionality and disability, is based on the concepts of the International Classification of Functioning, Disability and Health. It captures the level of functionality in 6 domains: cognition, mobility, self-care, interaction with others, day-to-day activities, and participation in society.(from 0 - no difficulty to 4 - extreme difficulty or can not do). A higher score corresponds to a worse level of functionality. It is a simple and easy to apply (5 minutes) measure, being valid and reliable. It will be applied to people with CRD and their informal carers.
Zarit Burden Interview (ZBI-22) | Task 2 and 3 (baseline)
  The ZBI-22 is used to assess the perception of informal carers regarding the impact of the disease on their lives, health and well-being, and social and financial life. It is composed of 22 assertions, scored from 0 (never) to 4 (almost always). The total score ranges from 0 to 88 and a higher score indicates greater burden. It is used worlwide in different contexts. It will be applied to informal carers of people with CRD.
Positive Aspects of Caregiving (PAC) | Task 2 and 3 (baseline)
  The PAC scale reflects the positive aspects of caring for someone, as an informal/family carer,being an adaptation of the Caregiver Satisfaction Scale. It includes 11 items, scored from 1 (disagree a lot) to 5 (agree a lot). The score varies from 11 to 55, and a higher score corresponds to a better perception of the experience as an informal/family carer. It has been used in different contexts and has good measurement properties. It will be applied to informal carers of people with CRD.
European Health Literacy Survey - 47 items (HLS-EU-Q47) | Task 2 and 3 (baseline)
  The HLS-EU-Q47 was developed to assess health literacy considering the current definition of this concept. It consists of 47 items, integrating 3 domains (health care, health promotion and disease prevention) and 4 levels of information processing (access, understanding, evaluation and use). The analysis of health literacy is performed in 12 sub-indexes, which are scored on a 4-point scale (very difficult, difficult, easy, very easy). A higher score corresponds to better health literacy. It will be applied to informal carers of people with CRD.
Carer Support Needs Assessment Tool (CSNAT) | Task 2 and 3 (baseline)
  The CNSAT was developed to assess the needs of informal carers of people with cancer in the terminal phase. This measure has 5 phases: 1. introduction of the instrument; 2. completion of the instrument in its 15 domains; 3. an interview/guided conversation between the carer and the health professional, in which the needs of the carer are identified and prioritized; 4. adaptation solutions to the priorities; 5. review of the results. The process is then repeated at an agreed moment. It is valid and sensitive to change. It will be applied to informal carers of people with CRD and used as content validity to the instrument that will be developed in this project.
Qualitative data: interviews | Task 2 and 3 (baseline)
  People with CRD and their informal carers, as well as health professionals, may participate in a interview in order to identify, understand and prioritize the needs of informal carers of people with CRD. Data from the interviews will be compared.
  For the development of the new instrument, individual cognitive interviews will be conducted with informal carers of people with CRD to refine its final version.
Social connectedness and care-related questions | Task 2 and 3 (baseline)
  People with CRD and their informal carers: Geographical proximity to most of the social network; Social participation; Number of people providing informal care; Type of support received/provided; Relationship with the care provider/recipient; How good is the relationship with the care provider/recipient; Do you live with the care provider/recipient; Hours spent receiving/providing informal care per week; Frequency of informal care received/provided per week; Duration of informal care received/provided; Do you provide care to someone;
  People with CRD: Formal/informal care; Types of formal care; Hours spent receiving formal care per week; Satisfaction with informal care received
  Informal Carers of people with CRD: Recognised informal care status; Number of people providing care for; Impact on job/work due to caring for someone; Impact on sleep due to caring for someone
Brief Physical Activity Assessment Tool (BPAAT) | Task 2 and 3 (baseline)
  The BPAAT was developed for healthcare professionals to identify inactive people in primary health care, identifying people who are sufficiently or insufficiently active. It consists of 2 questions: one on vigorous physical activity and the other on moderate physical activity, during an usual week. A total score ranges from 0 to 8 ( a score from 0 to 3 - not sufficiently active; and a score ≥4 - sufficiently active). It is easy to apply (5 minutes) and it is a valid and reliable measure, including for people with COPD. It will be applied to people with CRD and their informal carers.

OTHER OUTCOMES:
Sociodemographic data | Task 2 and 3 (baseline)
  People with CRD: Sex; Age; Year of birth; Level of education; Occupation; Type of employment contract; Marital status; Municipality; Area of residence; Home ownership; Type of housing; Physical modifications to the house due to the CRD; Religious affiliation; Race;Socio-economic status (gross monthly income)
  Informal carers of people with CRD: Sex; Age; Year of birth; Level of education; Occupation; Type of employment contract; Marital status; Municipality; Area of residence; Home ownership; Type of housing; Religious affiliation; Race;Socio-economic status (gross monthly income)
  Health professionals: Sex; Age; Year of birth; Level of education; Specialisation
Clinical data | Task 2 and 3 (baseline)
  People with CRD: Cognitive status (6-item cognitive impairment test); Diagnosis; Year of diagnosis; Disease stage; Lung function; Smoking status; Long-term Oxygen Therapy; Non-invasive ventilation; Comorbidities; Medication; Healthcare utilisation in the previous year; Number of exacerbations in previous year; Number of falls; Mobility aids
  Informal carerss of people with CRD: Smoking status; Comorbidities; Medication; Healthcare utilisation in the previous year; Number of falls
Anthropometric data | Task 2 and 3 (baseline)
  People with CRD and their informal carers: height (meters); weight (Kg); Body mass index (kg/m^2)
Contact with people with CRD | Task 2 (baseline)
  Health professionals: Duration of contact with peple with CRD in clinical practice

CONTACTS AND LOCATIONS:
Overall Officials: Alda S Marques, PhD, Principal Investigator — School of Health Sciences of the University of Aveiro (ESSUA)
Locations (1):
- University of Aveiro, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2019 Chronic Respiratory Diseases Collaborators. Global burden of chronic respiratory diseases and risk factors, 1990-2019: an update from the Global Burden of Disease Study 2019. EClinicalMedicine. 2023 May;59:101936. doi: 10.1016/j.eclinm.2023.101936. PMID 37229504
- [Background] Kaptain RJ, Helle T, Patomella AH, Weinreich UM, Kottorp A. New Insights into Activities of Daily Living Performance in Chronic Obstructive Pulmonary Disease. Int J Chron Obstruct Pulmon Dis. 2021 Jan 7;16:1-12. doi: 10.2147/COPD.S264365. eCollection 2021. PMID 33447024
- [Background] Nakazawa A, Cox NS, Holland AE. Current best practice in rehabilitation in interstitial lung disease. Ther Adv Respir Dis. 2017 Feb;11(2):115-128. doi: 10.1177/1753465816676048. Epub 2016 Nov 15. PMID 28150539
- [Background] Lee JYT, Tikellis G, Corte TJ, Goh NS, Keir GJ, Spencer L, Sandford D, Khor YH, Glaspole I, Price J, Hey-Cunningham AJ, Maloney J, Teoh AKY, Watson AL, Holland AE. The supportive care needs of people living with pulmonary fibrosis and their caregivers: a systematic review. Eur Respir Rev. 2020 Apr 29;29(156):190125. doi: 10.1183/16000617.0125-2019. Print 2020 Jun 30. PMID 32350085
- [Background] Pena-Longobardo LM, Oliva-Moreno J, Hidalgo-Vega A, Miravitlles M. Economic valuation and determinants of informal care to disabled people with Chronic Obstructive Pulmonary Disease (COPD). BMC Health Serv Res. 2015 Mar 15;15:101. doi: 10.1186/s12913-015-0759-6. PMID 25889556
- [Background] Dzingina MD, Reilly CC, Bausewein C, Jolley CJ, Moxham J, McCrone P, Higginson IJ, Yi D. Variations in the cost of formal and informal health care for patients with advanced chronic disease and refractory breathlessness: A cross-sectional secondary analysis. Palliat Med. 2017 Apr;31(4):369-377. doi: 10.1177/0269216317690994. Epub 2017 Feb 13. PMID 28190370
- [Background] Macdonald MT, Lang A, Storch J, Stevenson L, Barber T, Iaboni K, Donaldson S. Examining markers of safety in homecare using the international classification for patient safety. BMC Health Serv Res. 2013 May 24;13:191. doi: 10.1186/1472-6963-13-191. PMID 23705841
- [Background] Cruz J, Marques A, Figueiredo D. Impacts of COPD on family carers and supportive interventions: a narrative review. Health Soc Care Community. 2017 Jan;25(1):11-25. doi: 10.1111/hsc.12292. Epub 2015 Oct 26. PMID 26499310
- [Background] Trivedi RB, Bryson CL, Udris E, Au DH. The influence of informal caregivers on adherence in COPD patients. Ann Behav Med. 2012 Aug;44(1):66-72. doi: 10.1007/s12160-012-9355-8. PMID 22422104
- [Background] Kong YL, Anis-Syakira J, Jawahir S, R'ong Tan Y, Rahman NHA, Tan EH. Factors associated with informal caregiving and its effects on health, work, and social activities of adult informal caregivers in Malaysia: findings from the National Health and Morbidity Survey 2019. BMC Public Health. 2021 Jun 1;21(1):1033. doi: 10.1186/s12889-021-11022-1. PMID 34074275
- [Background] Terwee CB, Prinsen CAC, Chiarotto A, Westerman MJ, Patrick DL, Alonso J, Bouter LM, de Vet HCW, Mokkink LB. COSMIN methodology for evaluating the content validity of patient-reported outcome measures: a Delphi study. Qual Life Res. 2018 May;27(5):1159-1170. doi: 10.1007/s11136-018-1829-0. Epub 2018 Mar 17. PMID 29550964
- [Background] Health measurement scales: a practical guide to their development and use (5th edition). Aust N Z J Public Health. 2016 Jun;40(3):294-5. doi: 10.1111/1753-6405.12484. No abstract available. PMID 27242256
- [Background] Apostolo JLA, Paiva DDS, Silva RCGD, Santos EJFD, Schultz TJ. Adaptation and validation into Portuguese language of the six-item cognitive impairment test (6CIT). Aging Ment Health. 2018 Sep;22(9):1184-1189. doi: 10.1080/13607863.2017.1348473. Epub 2017 Jul 25. PMID 28741373
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Tomaszewski EL, Atkinson MJ, Janson C, Karlsson N, Make B, Price D, Reddel HK, Vogelmeier CF, Mullerova H, Jones PW; NOVELTY Scientific Community; NOVELTY study investigators. Chronic Airways Assessment Test: psychometric properties in patients with asthma and/or COPD. Respir Res. 2023 Apr 8;24(1):106. doi: 10.1186/s12931-023-02394-6. PMID 37031164
- [Background] Patel AS, Siegert RJ, Brignall K, Gordon P, Steer S, Desai SR, Maher TM, Renzoni EA, Wells AU, Higginson IJ, Birring SS. The development and validation of the King's Brief Interstitial Lung Disease (K-BILD) health status questionnaire. Thorax. 2012 Sep;67(9):804-10. doi: 10.1136/thoraxjnl-2012-201581. Epub 2012 May 3. PMID 22555278
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Pais-Ribeiro J, Silva I, Ferreira T, Martins A, Meneses R, Baltar M. Validation study of a Portuguese version of the Hospital Anxiety and Depression Scale. Psychol Health Med. 2007 Mar;12(2):225-35; quiz 235-7. doi: 10.1080/13548500500524088. English, Portuguese. PMID 17365902
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Lubben J, Blozik E, Gillmann G, Iliffe S, von Renteln Kruse W, Beck JC, Stuck AE. Performance of an abbreviated version of the Lubben Social Network Scale among three European community-dwelling older adult populations. Gerontologist. 2006 Aug;46(4):503-13. doi: 10.1093/geront/46.4.503. PMID 16921004
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Kusier AO, Folker AP. The Satisfaction with Life Scale: Philosophical Foundation and Practical Limitations. Health Care Anal. 2021 Mar;29(1):21-38. doi: 10.1007/s10728-020-00420-y. Epub 2021 Jan 2. PMID 33386535
- [Background] Lee Y, Li L. Evaluating the Positive Experience of Caregiving: A Systematic Review of the Positive Aspects of Caregiving Scale. Gerontologist. 2022 Oct 19;62(9):e493-e507. doi: 10.1093/geront/gnab092. PMID 34216215
- [Background] Archbold PG, Stewart BJ, Greenlick MR, Harvath T. Mutuality and preparedness as predictors of caregiver role strain. Res Nurs Health. 1990 Dec;13(6):375-84. doi: 10.1002/nur.4770130605. PMID 2270302
- [Background] Sorensen K, Pelikan JM, Rothlin F, Ganahl K, Slonska Z, Doyle G, Fullam J, Kondilis B, Agrafiotis D, Uiters E, Falcon M, Mensing M, Tchamov K, van den Broucke S, Brand H; HLS-EU Consortium. Health literacy in Europe: comparative results of the European health literacy survey (HLS-EU). Eur J Public Health. 2015 Dec;25(6):1053-8. doi: 10.1093/eurpub/ckv043. Epub 2015 Apr 5. PMID 25843827
- [Background] Ewing G, Grande G; National Association for Hospice at Home. Development of a Carer Support Needs Assessment Tool (CSNAT) for end-of-life care practice at home: a qualitative study. Palliat Med. 2013 Mar;27(3):244-56. doi: 10.1177/0269216312440607. Epub 2012 Mar 26. PMID 22450160
- [Background] Cruz J, Jacome C, Oliveira A, Paixao C, Rebelo P, Flora S, Januario F, Valente C, Andrade L, Marques A. Construct validity of the brief physical activity assessment tool for clinical use in COPD. Clin Respir J. 2021 May;15(5):530-539. doi: 10.1111/crj.13333. Epub 2021 Feb 15. PMID 33484059
- See also: World Health Organization (WHO). The top 10 causes of death. World Health Organization 2020 — https://www.who.int/news-room/fact-sheets/detail/the-top-10-causes-of-death
- See also: Marques A, Goldstein RS. Living with chronic lung disease: The experiences and needs of patients and caregivers. Pulmonary Rehabilitation 2020:281. — https://www.taylorfrancis.com/chapters/edit/10.1201/9781351015592-29/living-chronic-lung-disease-experiences-needs-patients-caregivers-alda-marques-roger-goldstein
- See also: Eurocarers. Enabling carers to care: An EU strategy to support and empower informal carers. European Association working for carers 2023 — https://eurocarers.org/publications/enabling-carers-to-care/
- See also: World Health Organization. Measuring Health and Disability Manual for WHO Disability Assessment Schedule.; 2010 — https://www.who.int/publications/i/item/measuring-health-and-disability-manual-for-who-disability-assessment-schedule-(-whodas-2.0)